CLINICAL TRIAL: NCT03439618
Title: Comparison of Time-restricted Feeding and Continuous Feeding in Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qingdao University (Other)
Responsible Party: Principal Investigator, Bo Yao,phD, Clinician of intensive care unit, Principal Investigator, Qingdao University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YB201811
Record Dates: First submitted 2018-01-31; First posted 2018-02-20 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Feeding Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- continuous feeding (Other): The total amount of every days' Enteral Nutritional Suspension was fed at constant speed for 24h
  Interventions: Other: continuous feeding
- time-restricted feeding (Other): The total amount of every days' Enteral Nutritional Suspension was fed at constant speed for 6h (7:00-9:00,11:00-13:00,17:00-19:00).
  Interventions: Other: time-restricted feeding

INTERVENTIONS:
Other: time-restricted feeding — At the beginning, all enrolled patients were fed by continuous feeding. When the amount calorie of feeding enteral nutritional suspension increased to 80% target calorie (target calorie: 25kilocalorie/kg.d), the patients was randomly into continuous feeding and time-restricted feeding group. In continuous feeding group, the enteral nutritional suspension was fed at constant speed for 24h.In the time restricted feeding, feeding time should be at 7:00-9:00, 11:00-13:00 and 17:00-19:00 at constant feeding speed.
  Arms: time-restricted feeding
Other: continuous feeding — At the beginning, all enrolled patients were fed by continuous feeding. When the amount calorie of feeding enteral nutritional suspension increased to 80% target calorie (target calorie: 25kilocalorie/kg.d), the patients was randomly into continuous feeding and time-restricted feeding group.In the continuous feeding, the total amount of every days' Enteral Nutritional Suspension was fed at constant speed for 24h.
  Arms: continuous feeding

SUMMARY:
In the nutrition guideline (A.S.P.E.N guideline), there was no recommendation about the feeding type in enteral feeding of critically ill patients. Continuous feeding is the most popular feeding type in ICU because of its less nursing burden and reducing the aspiration incidence theoretically. However, some previous studies demonstrated that there were no complications differences between continuous and time-restricted feedings（such as intermittent feedings）.

In ICU, the disorder of protein synthesis is a universal problem and is associated with ICU acquired weakness. Time-restricted feeding is more physical than continuous feeding. In some animal researches, time-restricted feeding was proved to have a greater stimulatory effect on protein synthesis than continuous feeding. Besides of light, time-restricted feeding can may also adjust the biological rhythms. It is known that biological clocks could affect energy metabolism, emotion and so on. Until now, there are no enough clinical studies to prove the advantages in time-restricted feeding in ICU patients.So researchers designed the study to compare the time-restricted feeding and continuous feeding effect(especially protein synthesis) on ICU patients.

DETAILED DESCRIPTION:
Enteral nutrition support can be administered by continuous administration or by time-restricted administration in ICU. Continuous feeding is the most popular feeding schedule because of its less nursing burden and reducing the aspiration prevalence theoretically. However, previous studies demonstrated that there was no complications (diarrhea, distension, Ventilator associated pneumonia-VAP incidence, and so on) difference between these two feeding schedule. So in the nutrition guideline (A.S.P.E.N guideline), there was no recommendation about the feeding schedule. However, time-restricted feeding is more physical than continuous feeding. In ICU, the disorder of protein synthesis is a universal problem and is associated with ICU acquired weakness. In some animal researches, time-restricted feeding was proved to have a greater stimulatory effect on protein synthesis than continuous feeding.

Besides of light, time-restricted feeding can adjust the biological rhythms. It is known that biological clocks could affect energy metabolism, emotion and so on. In the "zi wu liu zhu" theory of traditional chinese medicine, feeding time should be at 7:00-9:00, 11:00-13:00 and 17:00-19:00. So researchers designed the study to compare the time-restricted feeding according to traditional chinese medicine and continuous feeding effect(especially protein synthesis) on ICU patients.

ELIGIBILITY:
Inclusion Criteria:

ICU patients asking for enteral nutrition by gastric tube

Exclusion Criteria:

Patients with gastrectomy; patients with enterectomy; patients with Gastrointestinal hemorrhage; patients with diabetes; patients with intestinal fistula

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2018-05-09 (Actual); Primary Completion 2021-05-08 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
nitrogen balance | at the time point of 10th feeding day
  it equal to Nitrogen intake minus Nitrogen output.Source of nitrogen intake is the enteral nutritional suspension, and the amount of nitrogen can be calculated according to the proportion of nitrogen in enteral nutritional suspension. Main nitrogen losses include urine and feces. The amount of nitrogen in urine and feces can be measured by clinical laboratory.

SECONDARY OUTCOMES:
delirium | up to 10 days
  it is disorders of the mental state and medical condition. It can be evaluated by The Confusion Assessment Method for the Intensive Care Unit (CAM-ICU).
Gastric residual volume | up to 10 days
  This index was to evaluate the feeding complications. Nurse can evaluate the volume by pumping the stomach tube with syringe to measure the gastric content amount.
diarrhea | up to 10 days
  This index was to evaluate the feeding complications. It is the condition of having at least three loose or liquid bowel movements each day.
Incidence of ventilator-associated pneumonia | up to 10 days
  This index was to evaluate the feeding complications. Ventilator-associated pneumonia (VAP) is a type of lung infection that occurs in people who are on mechanical ventilation breathing machines for at least 48 hours. The diagnosis of VAP varies among hospitals and providers but usually requires a new infiltrate on chest x-ray plus two or more other factors. These factors include temperature of >38 or <36 °C, a white blood cell count of >12 × 10^9/ml, purulent secretions from the airways in the lung, and/or reduction in gas exchange.
glucose fluctuation | up to 10 days
  This index was to evaluate the feeding complications. The glucose is measured at the 11:00, 15:00, 21:00, 1:00 and 5:00 five time points. The glucose fluctuation is the maximum glucose amount plus minimum glucose amount.
Albumin | up to 10 days
  Serum albumin is the main protein of human blood plasma. It can be measured by clinical laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: BO Yao, PHD, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The affiliated hospital of qingdao university, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Patel JJ, Rosenthal MD, Heyland DK. Intermittent versus continuous feeding in critically ill adults. Curr Opin Clin Nutr Metab Care. 2018 Mar;21(2):116-120. doi: 10.1097/MCO.0000000000000447. PMID 29232262
- [Result] Sunderram J, Sofou S, Kamisoglu K, Karantza V, Androulakis IP. Time-restricted feeding and the realignment of biological rhythms: translational opportunities and challenges. J Transl Med. 2014 Mar 28;12:79. doi: 10.1186/1479-5876-12-79. PMID 24674294
- [Result] McClave SA, Taylor BE, Martindale RG, Warren MM, Johnson DR, Braunschweig C, McCarthy MS, Davanos E, Rice TW, Cresci GA, Gervasio JM, Sacks GS, Roberts PR, Compher C; Society of Critical Care Medicine; American Society for Parenteral and Enteral Nutrition. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). JPEN J Parenter Enteral Nutr. 2016 Feb;40(2):159-211. doi: 10.1177/0148607115621863. No abstract available. PMID 26773077
- [Result] Tavares de Araujo VM, Gomes PC, Caporossi C. Enteral nutrition in critical patients; should the administration be continuous or intermittent? Nutr Hosp. 2014 Mar 1;29(3):563-7. doi: 10.3305/nh.2014.29.3.7169. PMID 24559000
- [Result] Chen YC. Critical analysis of the factors associated with enteral feeding in preventing VAP: a systematic review. J Chin Med Assoc. 2009 Apr;72(4):171-8. doi: 10.1016/S1726-4901(09)70049-8. PMID 19372071
- [Result] Marik PE. Feeding critically ill patients the right 'whey': thinking outside of the box. A personal view. Ann Intensive Care. 2015 Dec;5(1):51. doi: 10.1186/s13613-015-0051-2. Epub 2015 May 28. PMID 26055186
- [Result] Wang HB, Loh DH, Whittaker DS, Cutler T, Howland D, Colwell CS. Time-Restricted Feeding Improves Circadian Dysfunction as well as Motor Symptoms in the Q175 Mouse Model of Huntington's Disease. eNeuro. 2018 Jan 3;5(1):ENEURO.0431-17.2017. doi: 10.1523/ENEURO.0431-17.2017. eCollection 2018 Jan-Feb. PMID 29302618
- [Derived] Ren CJ, Yao B, Tuo M, Lin H, Wan XY, Pang XF. Comparison of sequential feeding and continuous feeding on the blood glucose of critically ill patients: a non-inferiority randomized controlled trial. Chin Med J (Engl). 2021 Jul 20;134(14):1695-1700. doi: 10.1097/CM9.0000000000001684. PMID 34397596